CLINICAL TRIAL: NCT02005978
Title: Incretin Effect and Gastrointestinally Mediated Glucose Disposal in Cranially Irradiated Patients With Acromegaly
Brief Title: Brain-gut Interaction in Irradiated Patients With Acromegaly
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Ulla Feldt-Rasmussen, Professor, chief physician, Rigshospitalet, Denmark
Other Study IDs: ACRO-INC-TME
Record Dates: First submitted 2013-11-18; First posted 2013-12-09 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Acromegaly1: Acromegalic patients treated with radiation therapy
- Healthy controls: Health controls matched for age, gender and BMI to the patients
- Acromegaly 2: Acromegalic patients treated with pituitary surgery

SUMMARY:
Acromegaly is caused by increased production of growth hormone (GH) from a usually benign pituitary tumor. The disease causes a number of complications including disturbances in glucose metabolism and about 25% of the patients develop diabetes. Most patients are cured upon surgery alone, but many require additional medical treatment, and in rare cases radiotherapy. A disadvantage of radiotherapy is a risk of radiation damage to nearby areas such as the hypothalamus. The true extent of irradiation induced hypothalamic dysfunction, however, remains uncertain.

Data have shown significant improvement and often normalization of glucose metabolism upon surgical cure from acromegaly, whereas data suggest that such improvement is less likely in patients receiving additional radiotherapy.

The hypothalamus is part of the so-called 'gut-brain axis', where gastrointestinal hormones through interaction with the hypothalamus plays a significant role in the regulation of appetite and glucose metabolism. Incretins are the most prominent gastrointestinal hormones involved, with the incretin-effect referring to food-induced insulin secretion, which in healthy subjects is responsible for up to 70% of the insulin response after oral glucose intake. The investigators hypothesize that radiation conditional influence of the hypothalamus may compromise the gut-brain activity and thereby affect the incretin-effect and gastrointestinal-mediated glucose disposal (GIGD; i.e. sum of all gastrointestinal-derived factors that contribute to glucose metabolism) in patients with acromegaly. The aim of the study is to investigate the long term effect of surgery with or without additional fractionated radiation therapy on glucose metabolism as assessed by incretin-effect and GIGD in acromegaly, in order to identify possible associations with treatment modality.

The study population include 24 acromegalic patients who have previously received (N=12) or did not receive (N=12) pituitary irradiation as part of their treatment, and 12 matched healthy controls.

DETAILED DESCRIPTION:
Acromegaly is caused by increased production of growth hormone (GH) from a usually benign pituitary tumor. The disease causes a number of complications including disturbances in glucose metabolism and about 25% of the patients develop diabetes. Most patients are cured upon surgery alone, but many require additional medical treatment, and in rare cases radiotherapy. A disadvantage of radiotherapy is a risk of radiation damage to nearby areas such as the hypothalamus. The true extent of irradiation induced hypothalamic dysfunction, however, remains uncertain.

Data have shown significant improvement and often normalization of glucose metabolism upon surgical cure from acromegaly, whereas data suggest that such improvement is less likely in patients receiving additional radiotherapy.

The hypothalamus is part of the so-called 'gut-brain axis', where gastrointestinal hormones through interaction with the hypothalamus plays a significant role in the regulation of appetite and glucose metabolism. Incretins are the most prominent gastrointestinal hormones involved, with the incretin-effect referring to food-induced insulin secretion, which in healthy subjects is responsible for up to 70% of the insulin response after oral glucose intake. The investigators hypothesize that radiation conditional influence of the hypothalamus may compromise the gut-brain activity and thereby affect the incretin-effect and gastrointestinal-mediated glucose disposal (GIGD; i.e. sum of all gastrointestinal-derived factors that contribute to glucose metabolism) in patients with acromegaly.

The aim of the study is to investigate the long term effect of surgery with or without additional fractionated radiation therapy on glucose metabolism as assessed by incretin-effect and GIGD in acromegaly, in order to identify possible associations with treatment modality.

Design: observational case-control study Participants: Acromegalic patients who have previously received (N=12) or did not receive (N=12) pituitary irradiation as part of their treatment, and 12 matched healthy controls.

Investigation: Extended oral glucose tolerance test (OGTT), followed by isoglycaemic intravenous glucose infusion (IGII) with concurrent measurement of plasma-glucose, -insulin, -C-peptide, -glucagon, glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic peptide (GIP) at fixed time-points.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of acromegaly, and treated at the department of Endocrinology, Copenhagen University Hospital, Rigshospitalet, Denmark (tertiary referral hospital)

Exclusion Criteria:

* Diabetes mellitus
* Pregnancy or breastfeeding
* Treatment with medications potentially influencing glucose metabolism, including thiazides and steroids (replacement therapy with hydrocortisone not included but matched for).
* Chronic or earlier events of acute pancreatitis
* Inflammatory bowel disease (Mb. Crohn/ulcerous colitis)
* Bowel resection or larger gastrointestinal surgical interventions
* Blood percent < 6.5 mmol/L

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acromegaly treated with radiation therapy or surgery
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Measure the incretin effect during glucose tolerance tests in acromegaly | one year
  Extended oral glucose tolerance test (OGTT), followed by isoglycaemic intravenous glucose infusion (IGII) with concurrent measurement of plasma-glucose, -insulin, -C-peptide, -glucagon, glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic peptide (GIP) at fixed time-points.

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Feldt-Rasmussen, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- National University Hospital, Department of Medical Endocrinology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jorgensen NT, Erichsen TM, Jorgensen MB, Idorn T, Feldt-Rasmussen B, Holst JJ, Feldt-Rasmussen U, Klose M. Glucose metabolism, gut-brain hormones, and acromegaly treatment: an explorative single centre descriptive analysis. Pituitary. 2023 Feb;26(1):152-163. doi: 10.1007/s11102-022-01297-x. Epub 2023 Jan 6. PMID 36609655